CLINICAL TRIAL: NCT00068185
Title: Interactions Between SERMs, Soy and Black Cohosh
Brief Title: A Study of the Pharmacokinetics of Black Cohosh
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution, study did not continue, funding stopped
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Heather Shaw, MD, Duke University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K08AT001315-01A1 (NIH)
Record Dates: First submitted 2003-09-09; First posted 2003-09-10 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Hot Flashes
Keywords: Black cohosh; Pharmacokinetics; Alternative therapies; Natural product
MeSH Terms: conditions — Hot Flashes | interventions — black cohosh root extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Black cohosh

SUMMARY:
Black cohosh is a natural supplement that has been used to treat and prevent menopausal symptoms. Remifemin is a standardized form of black cohosh. The purpose of this study is to determine the levels of components of black cohosh obtained in the blood of healthy women taking Remifemin.

DETAILED DESCRIPTION:
As per Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* No prior diagnosis of cancer other than non-melanoma skin cancer or carcinoma in-situ of the cervix
* No current prescription medication use
* Negative urine pregnancy test OR greater than age 50 with no menses for at least one year OR documented status post hysterectomy
* Competent to understand and sign informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2003-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather S Shaw, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States